CLINICAL TRIAL: NCT00371956
Title: Raloxifene for Prevention of Bone Loss in Postmenopausal Patients Receiving Chronic Corticosteroid Therapy: a Randomized Double-blind Placebo-controlled Study
Brief Title: Raloxifene for Prevention of Bone Loss in Postmenopausal Patients Receiving Chronic Corticosteroid Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: CC Mok, Tuen Mun Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HARECCTR0500058
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Osteoporosis
Keywords: raloxifene; estrogen; receptor; modulation; osteoporosis; steroid; Steroids
MeSH Terms: conditions — Osteoporosis | interventions — Raloxifene Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): raloxifene
  Interventions: Drug: raloxifene
- 2 (Placebo Comparator): placebo arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: raloxifene — 60mg/day
  Arms: 1
Drug: placebo — tab 1 daily
  Arms: 2

SUMMARY:
This study is a double-blind placebo-controlled trial evaluating the efficacy of raloxifene in the prevention of bone mineral density loss in patients receiving long term corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal patients with various chronic rheumatic diseases receiving chronic steroid therapy.
2. Stable disease for at least 6 months prior to study with a stable dose of steroid (prednisone <= 10 mg/day or equivalent).
3. Baseline bone mineral density (BMD) of the lumbar spine T score < -1.0.

Exclusion Criteria:

1. Patients with a history of thromboembolism.
2. Patients with positive antiphospholipid antibodies.
3. History of allergic reactions or intolerance to raloxifene or other SERMs.
4. Patients receiving bisphosphonates, parathyroid hormone, SERMs, anticonvulsants or anti-cytokine therapies within 6 months prior to study entry.
5. Patients with known bone disorders such as osteomalacia, renal osteodystrophy, and hyperparathyroidism.
6. Patients with abnormal uterine bleeding of unknown etiology.
7. Patients with serum creatinine level of >= 200 umol/L.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2006-09; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Bone turnover and bone mineral density | 12 months

SECONDARY OUTCOMES:
Fracture, safety | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: CC MOK, MD, FRCP, Principal Investigator — Tuen Mun Hospital Hong Kong
Locations (1):
- Tuen Mun Hospital, Hong Kong, China

REFERENCES:
- [Derived] Mok CC, Ying KY, To CH, Ho LY, Yu KL, Lee HK, Ma KM. Raloxifene for prevention of glucocorticoid-induced bone loss: a 12-month randomised double-blinded placebo-controlled trial. Ann Rheum Dis. 2011 May;70(5):778-84. doi: 10.1136/ard.2010.143453. Epub 2010 Dec 27. PMID 21187295